CLINICAL TRIAL: NCT01191788
Title: Group Cognitive Behavioral Therapy (CBT) For Depression in Clients With Alcohol and Other Drug (AOD) Disorders
Brief Title: Building Recovery By Improving Goals, Habits, and Thoughts
Acronym: BRIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Behavioral Health Services, Inc. (Industry); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01AA014699-03 (NIH); R01AA014699 (NIH)
Record Dates: First submitted 2010-06-29; First posted 2010-08-31 (Estimated); Results first posted 2012-06-25 (Estimated); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Depression; Substance Use
Keywords: Depression; Substance Use; Group Cognitive Behavioral Therapy
MeSH Terms: conditions — Depression; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group CBT (Experimental): Clients received up to 16 sessions of group CBT for depression
  Interventions: Behavioral: Group Cognitive Behavioral Therapy; Behavioral: Group CBT for Depression
- Comparison (Active Comparator): Treatment as Usual comparison condition
  Interventions: Behavioral: Group Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Group Cognitive Behavioral Therapy — 16 two hour sessions of group CBT
Behavioral: Group CBT for Depression — 16 of group CBT for depression delivered in 2 hour groups for up to 8 weeks by a trained substance abuse treatment counselor
  Arms: Group CBT

SUMMARY:
The investigators will investigate whether group Cognitive Behavioral Therapy (CBT) for depression, with alcohol and other drug (AOD) treatment counselors leading the groups, is effective and cost effective in treating depression. If so, it could substantially increase access to appropriate mental health care. 360 clients with Beck Depression Inventory-II scores > 17 who are being treated in a single public sector AOD treatment organization will receive one of two conditions: (1) usual care residential AOD treatment (UC); (2) usual care AOD residential treatment plus a 16-session course of group CBT delivered by trained AOD counselors (CBT). Data will be analyzed using an intent-to-treat model. The investigators will collect data on the service-level costs and health effects associated with UC and CBT, and will calculate the incremental cost per unit of depression and AOD improvement, compared to UC.

DETAILED DESCRIPTION:
Individuals with alcohol and other drug (AOD) disorders frequently suffer from depression, leading to reduced quality of life and poorer AOD treatment outcomes. Efficacious treatments for depression do exist and could improve outcomes; but national data suggest that fewer than 7% of people with co-occurring disorders who are in AOD treatment have received appropriate treatment. Group cognitive behavioral therapy (CBT) is an effective and inexpensive treatment for depression. We propose to investigate whether group CBT for depression, with AOD counselors leading the groups, is effective and cost effective in treating depression. If so, it could substantially increase access to appropriate mental health care.

We propose a 5-year quasi-experimental study with the following specific aims: Aim 1. To evaluate the effectiveness of group CBT for depression provided by AOD counselors in improving depressive symptoms and AOD outcomes, among clients being treated in public sector residential AOD treatment settings; Aim 2. To evaluate the cost-effectiveness of group CBT conducted by trained AOD counselors compared to usual care AOD treatment; Aim 3. To document the implementation of the intervention at each of the four sites, and to determine whether the AOD counselors are delivering the group CBT intervention with fidelity to the model, and whether treatment fidelity is a significant predictor of client outcomes.

We will enroll and follow 360 clients with Beck Depression Inventory-II (BDI-II) scores > 17 who are being treated in a single public sector AOD treatment organization at four residential sites in LA County. Subjects will receive one of two conditions: (1) usual care residential AOD treatment (UC); (2) usual care AOD residential treatment plus a 16-session course of group CBT delivered by trained AOD counselors (CBT). Subjects will complete: (1) a baseline interview; (2) a post-treatment interview (at the conclusion of the CBT treatment) and (3) a follow-up interview (3 months after CBT treatment ends). Data will be analyzed using an intent-to-treat model. We will collect data on the service-level costs and health effects associated with UC and CBT, and will calculate the incremental cost per unit of depression and AOD improvement, compared to UC. . The implementation analysis will involve two related sets of activities: (1) a series of key informant interviews to provide a context in which to understand intervention implementation and (2) an assessment of treatment fidelity and it's relationship to client outcomes.

ELIGIBILITY:
Inclusion Criteria:

* present for treatment at one of four participating sites during study period
* score BDI>17 at 2-4 weeks post-treatment entry

Exclusion Criteria:

* cognitive impairment (score of 11 or greater on short Blessed exam)
* screen positive for bipolar or schizophrenia
* non-English speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2006-08; Primary Completion 2009-07 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Watkins, MD, MSHS, Principal Investigator — RAND
Locations (1):
- Behavioral Health Services, Inc, Gardena, California, United States

REFERENCES:
- [Derived] Watkins KE, Hunter S, Hepner K, Paddock S, Zhou A, de la Cruz E. Group cognitive-behavioral therapy for clients with major depression in residential substance abuse treatment. Psychiatr Serv. 2012 Jun;63(6):608-11. doi: 10.1176/appi.ps.201100201. PMID 22638007
- [Derived] Hunter SB, Witkiewitz K, Watkins KE, Paddock SM, Hepner KA. The moderating effects of group cognitive-behavioral therapy for depression among substance users. Psychol Addict Behav. 2012 Dec;26(4):906-16. doi: 10.1037/a0028158. Epub 2012 May 7. PMID 22564202
- [Derived] Watkins KE, Hunter SB, Hepner KA, Paddock SM, de la Cruz E, Zhou AJ, Gilmore J. An effectiveness trial of group cognitive behavioral therapy for patients with persistent depressive symptoms in substance abuse treatment. Arch Gen Psychiatry. 2011 Jun;68(6):577-84. doi: 10.1001/archgenpsychiatry.2011.53. PMID 21646576

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group CBT | Comparison
Started | 140 | 159
Completed | 119 (Completed 3-month followup) | 137 (Completed 3-month followup)
Not Completed | 21 | 22
Not completed — Lost to Follow-up | 21 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group CBT | Comparison | Total
Number analyzed (Participants) | 140 | 159 | 299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 139 | 159 | 298
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.31 (10.08) | 37.04 (10.53) | 36.23 (10.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 74 | 144
  Male | 70 | 85 | 155
Region of Enrollment [Number; unit: participants]
  United States | 140 | 159 | 299

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms as Measured by the Beck Depression Inventory II
Description: The Beck Depression Inventory II (BDI-II) is a 21 question, self-administered measure of depressive symptoms. Scores range from 0 - 63, with higher scores indicating more severe depressive symptoms.
Time Frame: 3 Months Post Treatment
Measure: Mean (Standard Deviation); unit: BDI-II score
Groups:
- Group CBT: Usual care + BRIGHT intervention. The BRIGHT intervention included 16 two-hour group sessions of CBT for depression.
- Comparison: Usual care
Arm/Group | Group CBT | Comparison
Number analyzed (Participants) | 120 | 140
BDI-II score | 14.83 (11.23) | 21.82 (12.74)

2. Secondary Outcome: Mental Health Functioning as Measured by SF-12 MCS.
Description: The SF-12 is a 12 question, self-administered measure of general health functioning. The SF-12 outputs a mental health summary score (MCS), which ranges from 0 to 100, with higher scores indicating better mental health functioning. MCS scores are standardized such that mean = 50 and SD = 10 in the general U.S. population.
Time Frame: 3 Months Post Treatment
Measure: Mean (Standard Deviation); unit: SF-12 score
Arm/Group | Group CBT | Comparison
Number analyzed (Participants) | 120 | 140
SF-12 score | 44.71 (11.34) | 38.44 (11.89)

ADVERSE EVENTS:
Arm/Group | Group CBT | Comparison
Serious Adverse Events (participants affected / at risk) | 0/140 | 0/159
Other Adverse Events (participants affected / at risk) | 0/140 | 0/159

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes